CLINICAL TRIAL: NCT05682469
Title: Effects and Mechanism of the Fully Immersive Virtual Reality Cognitive Training Based on Leisure Activities: Cognitive, Daily Function, Quality of Life, Metabolic Biomarkers, and Electroencephalography
Brief Title: Effects and Mechanism of the Fully Immersive Virtual Reality Cognitive Training Based on Leisure Activities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202102478B0
Record Dates: First submitted 2022-12-24; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: MCI; SCD
Keywords: Mild cognitive impairment; Subjective cognitive decline; Combination therapy; Virtual reality; Cognitive training; Leisure activities
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): VR cognitive training receives eight gardening activities. The cognitive elements including attention, working memory, processing speed, and executive function incorporated training.
  Interventions: Behavioral: VR cognitive training
- control group (Active Comparator): The control group is performing traditional cognitive training program.
  Interventions: Behavioral: Traditional cognitive training

INTERVENTIONS:
Behavioral: VR cognitive training — All participants will receive trainings for 60 minutes per day, two days per week for 16 sessions.
  All participants will receive one immersive leisure-based VR cognitive training for 40 minutes. VR cognitive training receives four gardening activities.
  The cognitive elements including attention, working memory, processing speed, and executive function incorporated training.
  Arms: VR group
Behavioral: Traditional cognitive training — All participants will receive trainings for 60 minutes per day, two days per week for 16 sessions.
  The control group is performing traditional cognitive training program.
  Arms: control group

SUMMARY:
The aim of this study is to identify the effects of the immersive leisure-based VR cognitive training, and compare the intervention effects for elderly with MCI and SCD. The investigators anticipate the VR training can facilitate cognitive function, daily function, quality of life. The investigators anticipated the metabolic biomarkers, mechanism, and brain activities will be found. The significance of this study is identifying the effect of immersive leisure-based VR cognitive training, and confirming the metabolic biomarkers and brain activities. It could improve the accuracy of identification, prevent the progression to dementia, and lead the field of technological assistance to new opportunities for training.

ELIGIBILITY:
Inclusion Criteria:

-

MCI Inclusion Criteria:

age>=60 able to follow instruction MoCA<26 Scores on cognitive tests for individuals with MCI are 1 to 1.5 standard deviations below the mean for their age and education matched peers on culturally

SCD Inclusion Criteria:

age>=60 ECog-12 score >1 MoCA>=26; does not conform the standards of MCI and dementia

Exclusion Criteria:

- dizziness or epilepsy history; neurological or other orthopedic diseases with neurological or other orthopedic diseases unstable physical condition of VR cognitive training Recent psychiatric diagnosis, such as depression

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change scores of the Montreal Cognitive Assessment (MoCA). | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Wechsler Memory Scale (WMS) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  including Faces Recognition (total scale=48), Verbal Paired Associates (total scale = 32), Word Lists (total scale = 48), and Spatial Span (total scale=32) will be used to assess the immediate, delayed, and working memory tests. For each subtest, a higher number indicates better performance in memory function. The raw score of subtests will also be transferred to standardized Z scores and summed to represent an index of general memory function.
Change scores of Stroop test | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. The time to complete the task will be calculated for each condition
Change scores of Color trials test | baseline, after the intervention eight weeks, and at 3-month follow-up.
  For Part 1, the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2, the respondent rapidly connects numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.
Change scores of Wechsler Adult Intelligence Scale; WAIS | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The digit symbol test involves a key consisting of the numbers 1-9, each paired with a unique, easy-to-draw symbol such as a "V", "+" or ">".
  Matrix Reasoning
  This is a nonverbal reasoning task in which individuals are asked to identify patterns in designs. This subtest measures:
  * non-verbal reasoning skills
  * broad visual intelligence
  * perceptual organization skills
Change scores of the short (12-item) form of the Everyday Cognition Scale (ECog-12) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The short (12-item) form of the Everyday Cognition Scale (ECog-12), which was developed as an informant-rated report of cognitively mediated functional abilities in older adults. The ECog-12 asks participants to rate their current ability to perform cognitively mediated daily tasks related to everyday memory, language, visuospatial abilities, and executive functions compared with their ability to do the same task 10 years ago. Items are rated on a scale of 1-4, with 1 = Better or no change and 4 = Consistently much worse. The global, executive, and memory ECog-12 sub-domain scores were generated by averaging over the component items (sum of items/number of items) to maintain a range of 1 to 4 (with higher scores reflecting greater self-reported SCD).
Change scores of Amsterdam Instrumental Activity of Daily Living,A-IADL | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Amsterdam Instrumental Activity of Daily Living (A-IADL) is an adaptive and computerized questionnaire designed to assess impairments in instrumental activities of daily living (IADL) in (early) dementia. The questionnaire is completed by a caregiver, such as a relative or friend.
  Each item has a 5-point scale response option (scored 0-4). The scoring of the Amsterdam Instrumental Activity of Daily Living is calculated using item response theory .Lower scores indicating poorer performance.
Change scores of Taiwan Performance-based IADL; TPIADL | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The TPIADL was designed to assess IADL ability in five domains: communication, finance, cooking, shopping and medicine use. To allow culture- and lifestyle-specific measurement, actual and simulated everyday objects were employed as stimulus materials.
  To develop more easily comprehensible stimuli materials, pictorial representations of a telephone directory and medication directions were used in the communication and medicine use tasks. Performance-based tasks were time-limited to 30 seconds, and the scoring reflected the level of efficiency in terms of the cognitive processing speed. The score for each task ranged from 1 to 3: 1 -completed without error and within 30 seconds; 2 -erroneous response within the time limit but corrected after a verbal cue; and 3 -not completed with errors within the time limit and unable to correct even following a verbal cue. The total score ranged from 5 to 15, with a higher score indicating a poorer performance in IADL.
Change scores of the World Health Organization Quality of Life-Old(WHOQOL-OLD) Taiwan Version | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The World Health Organization Quality of Life-Old questionnaires demonstrate acceptable psychometric performance in a convenience sample of Taiwan older people. It are valuable measures of Quality of Life-Old for use with older people.Time frame for assessment is the past two weeks.
  The items are distributed into 4 domains (physical; psychological, social and environmental health) and 25 facets.
Change scores of WHOQOL-bref Taiwan Version | baseline, after the intervention eight weeks, and at 3-month follow-up.
  As with the standard WHOQOL-BREF questionnaires the WHOQOL-BREF Taiwan version was simplified from the WHOQOL long form for Taiwan. For the purpose of cross-cultural comparison, the first 26 items were the same as the standard WHOQOL-BREF, which was developed from global studies. In addition to the 26 items, we applied the psychometric criteria proposed by the WHOQOL Group to select two more items from each of the two new facets to form the WHOQOL-BREF Taiwan version using data from the same 1,068 subjects. The selection process used for national items is described in the Results section. Thus, the WHOQOL-BREF Taiwan version contains 28 items classified into the same four domains as the standard WHOQOL-BREF. The scale administration and scoring procedures are the same as for the WHOQOL long form except that the facet score is based on only one item.
Change scores of Geriatric Depression Scale,GDS | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Geriatric Depression Scale (GDS) is a screening test originally developed by J.A. Yesavage and colleagues in 1982 that is used to identify symptoms of depression in older adults. The scale is a 30-item, self-report instrument that uses a "Yes/No" format.
Change scores of The Chinese Aging Well Profile (CAWP) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  It comprised eight open-ended questions focusing on the meaning and interpretation of 'subjective well-being', e.g., 'Can participants tell me what the important contributors to your well-being are?', 'Can participants describe the important elements in your life that make you feel happy?', 'Can participants describe the important elements in your life that participants dislike?' and 'What does well-being personally mean to participants?' To adapt the Aging Well Profile for a Chinese population in Taiwan was secured. It was agreed that the new version would be called the Chinese Aging Well Profile (CAWP).